CLINICAL TRIAL: NCT05049356
Title: Associated Symptoms, Underlying Mechanisms and Parental Factors of Child Psychiatric Disorders With Focus on Severe Irritability.
Brief Title: Symptoms and Mechanisms of Child Psychiatric Disorders
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: Linkoeping University (Other Government); Lovisenberg Diakonale Hospital (Other)
Responsible Party: Principal Investigator, Pål Zeiner, Head of Child Psychiatric Research, Oslo University Hospital
Other Study IDs: 2017/135
Record Dates: First submitted 2021-06-17; First posted 2021-09-20 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Disruptive Mood Dysregulation Disorder; Attention Deficit Hyperactivity Disorder; Oppositional Defiant Disorder; Severe Irritability; Child Psychiatric Disorders
Keywords: Neuropsychology; Neurocognition; Executive function; Social cognition; Mentalization; Affect recognition; Stress; Cortisol; Parental Stress; Attachment; Behavior symptoms; Emotion symptoms
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Oppositional Defiant Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Hair Cortisol Concentrations
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children referred to outpatient clinic: Diagnostic interview (Schedule for Affective Disorders and Schizophrenia (K-SADS) cf. Diagnostic and Statistical Manual of Mental Disorders (DSM-5)) with parents. Diagnostic groups/cohorts (e.g., DMDD, ADHD, Oppositional Defiant Disorder) will be based on the diagnoses given cf. K-SADS.
- Typical developing children and their parent(s): Norm values on hair cortisol data will be obtained from typical developing children and their parent(s) by the same procedure as described under Outcome measure(s), 21. Stress Response by Cortisol levels.

SUMMARY:
In this study the investigators will examine psychiatric symptoms, central neurocognitive functions, parental stress and attachment styles, and biological factors that can give new knowledge about some of the mechanisms present in children referred to outpatient psychiatric clinics. A specific focus will be given to children suffering from severe irritability.

DETAILED DESCRIPTION:
In this study the investigators will examine psychiatric symptoms, central neurocognitive functions, parental stress and attachment styles, and biological factors that can give new knowledge about some of the mechanisms present in children referred to outpatient psychiatric service. A specific focus will be given to children suffering from severe irritability making problems at home, in school, and/or with peers.

Disruptive Mood Dysregulation Disorder (DMDD) is characterized by chronic and severe irritability and anger in children. DMDD understood as severe or clinical irritability can be regarded as laying above a certain threshold on a irritability continuum. Due to DMDD being a relatively new and debated diagnosis there is an urgent need to gain better understanding of the underlying mechanisms of severe irritability in children.

This study will explore emotion and behavior symptoms, neuropsychological functions (including social perception), perceived parental stress and attachment styles, and cortisol levels of children and their mothers, in children referred to outpatient psychiatric service including children with severe irritability. Parents of children 6 to 12 years will be informed and asked to participate.

The work on severe irritability will be divided into six main areas:

1. Severe irritability in a Norwegian clinical population: prevalence, comorbidity and associated difficulties
2. Social and emotional understanding in severe irritability in children
3. Executive function in severe irritability in children
4. Stress response in severe irritability in children
5. Parental stress and attachment style in parents of severe irritability in children
6. DMDD: An affective or conduct disorder? Comparing anxiety and depressive symptoms

ELIGIBILITY:
Inclusion Criteria:

* Referred to outpatient psychiatric service
* Intelligence quotient (IQ) within normal range
* Child and parents: Good enough understanding of Norwegian language to give valid answers in interview and tests.
* Clarified care situation

Exclusion Criteria:

* IQ below normal range
* Child and parents: Not good enough understanding of Norwegian language to give valid answers in interview and tests
* Unclarified care situation

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Parents of children referred to outpatient psychiatric service (The Department of Child and Adolescent Psychiatry at Oslo University Hospital, and Nic Waals Institute at Lovisenberg Hospital) will be informed about the study and asked to participate.
Sampling Method: Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-08-09 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Social Perception by task performance: Affect Recognition | Baseline
  Affect Recognition, a subtest from the Developmental Neuropsychological Assessment (NEPSY®) Second Edition, will be used to measure facial affect recognition. In brief, higher scores means better recognition ability and vice versa:
  Total raw score:
  * 6 years old children: 4 (minimum) - 25 (maximum).
  * 7-12 years old children: 12 (min.) - 35 (max.).
  Raw scores are converted to scaled scores by Pearson's NEPSY-2 machine based scoring tool. Converted scaled scores have a mean of 10, a standard deviation of 3, and a range from 1-19.
Social Perception by task performance: Theory of Mind | Baseline
  Theory of Mind, a subtest from the NEPSY® Second Edition, will be used to measure the ability to understand that others have different thoughts, feelings and experiences than oneself. In brief, higher scores means better theory of mind ability and vice versa:
  Total raw score for 6-12 years old children: 0 (min.) - 28 (max.). Total Verbal raw score: 0 (min.) - 22 (max.). Raw scores are converted to percentiles* by Pearson's NEPSY-2 machine based scoring tool.
  *For scores with nonnormal distributions (i.e., underlying distribution were highly skewed), raw scores are converted to percentile ranks (instead of scaled scores).
Executive function by task performance: Verbal Working Memory | Baseline
  Word List Interference, a subtest from the NEPSY® Second Edition, will be used to measure Verbal Memory Span and Verbal Working Memory which are important executive functions.
  Scores for 7 to 12 years old children (not applicable to 6 years old):
  1. Repetition (WIRP)Total Score: 0 (min.) - 20 (max.).
  2. Recall (WIRC) Total Score: 0 (min.) - 40 (max.).
  Raw scores are converted to scaled scores* by Pearson's NEPSY-2 machine based scoring tool. Lower vs. higher scores on WIRP or WIRC means more limited vs. better Verbal Memory Span or Verbal Working Memory, respectively.
  *Converted scaled scores have a mean of 10, a standard deviation of 3, and a range from 1-19.
Executive function by task performance: Inhibitory Control | Baseline
  Inhibition, a subtests from the NEPSY® Second Edition, will be used to measure Inhibitory Control which is an important executive function. Scaled scores are calculated by Pearson's NEPSY-2 machine based scoring tool.
  In brief, a low Inhibition-Inhibition Combined Scaled Score* indicate poor Inhibitory Control, and a low Inhibition-Switching Combined Scaled Score* indicate poor Inhibitory Control and Cognitive Flexibility.
  The Inhibition-Inhibition Combined Scaled Score integrates error rate and time (i.e., raw score Inhibition-Inhibition Total Errors and Completion Time) with an emphasis on accuracy of performance over speed. .
  *Converted scaled scores have a mean of 10, a standard deviation of 3, and a range from 1-19.
Executive function by task performance: Cognitive Flexibility | Baseline
  Inhibition, a subtests from the NEPSY® Second Edition, will be used to measure Inhibitory Control and Cognitive Flexibility which are important executive functions. Scaled scores are calculated by Pearson's NEPSY-2 machine based scoring tool.
  In brief, a low Inhibition-Switching Combined Scaled Score* indicate poor Inhibitory Control and Cognitive Flexibility.
  The Inhibition-Switching Combined Scaled Score integrates error rates and time (i.e., raw score Inhibition-Switching Total Errors Completion Time) with more weight given on accuracy than speed.
  *Converted scaled scores have a mean of 10, a standard deviation of 3, and a range from 1-19.
Executive function by task performance: non-verbal Cognitive Flexibility | Baseline
  Design Fluency, a subtests from the NEPSY® Second Edition, will be used to measure Executive Function including non-verbal Cognitive Flexibility.
  Total raw score for 6 to 12 years old children: 0 (min.) - 70 (max.). Raw scores are converted to scaled scores* by Pearson's NEPSY-2 machine based scoring tool.
  In brief, higher scores scores means better non-verbal Cognitive Flexibility and Executive Function, and vice versa.
  *Converted scaled scores have a mean of 10, a standard deviation of 3, and a range from 1-19.
Executive function by report: Inhibitory control | Baseline
  Inhibitory control will be measured using the Behavior Rating Inventory of Executive Function, Second Edition (BRIEF-2; parent- and teacher-report) Inhibit Index. Items are converted from BRIEF to BRIEF-2 (cf. BRIEF-2 does not include additional items). Raw scores are calculated to t-scores according to the Psychological Assessment Resources' (PAR) BRIEF-2 manual. Higher scores mean worse ability to control impulses. T Scores ≥ 65 are regarded as in the clinical range.
  References:
  Gioia, G. A., Isquith, P. K., Guy, S. C., & Kenworthy, L. (2000). Behavior rating inventory of executive function professional manual. Odessa: FL: Psychological Assessment Resources.
  Gioia, G. A., Isquith, P. K., Guy, S. C., & Kenworthy, L. (2015). Behavior Rating Inventory of Executive Function®, Second Edition (BRIEF®2). Lutz, FL: PAR Inc.
Executive function by report: Cognitive flexibility | Baseline
  Cognitive flexibility (e.g., the ability to tolerate change and switch or alternate attention) will be measured using the BRIEF-2's Shift Index. Items are converted from BRIEF to BRIEF-2. Raw scores are calculated to t-scores according to the PAR BRIEF-2 manual. Higher scores mean worse ability to tolerate change and switch or alternate attention. T Scores ≥ 65 are regarded as in the clinical range.
Executive function by report: Emotional Control | Baseline
  Emotional control will be measured using the BRIEF-2's Emotional Control Index. Items are converted from BRIEF to BRIEF-2. Raw scores are calculated to t-scores according to the PAR BRIEF-2 manual. Higher scores means worse emotional control. T Scores ≥ 65 are regarded as in the clinical range.
Executive function by report: Initiate | Baseline
  The ability to begin an activity and to independently generate ideas or problem-solving strategies will be measured using the BRIEF-2's Initiate Index. Items are converted from BRIEF to BRIEF-2. Raw scores are calculated to t-scores according to the PAR BRIEF-2 manual. Higher scores means worse ability to initiate actions. T Scores ≥ 65 are regarded as in the clinical range.
Executive function by report: Working Memory | Baseline
  Working memory capacity will be measured using the BRIEF-2's Working Memory Index. Items are converted from BRIEF to BRIEF-2. Raw scores are calculated to t-scores according to the PAR BRIEF-2 manual. Higher scores means worse working memory. T Scores ≥ 65 are regarded as in the clinical range.
Executive function by report: Plan/Organize | Baseline
  Ability to plan/organize will be measured using the BRIEF-2's Plan/Organize Index. Items are converted from BRIEF to BRIEF-2. Raw scores are calculated to t-scores according to the PAR BRIEF-2 manual. Higher scores means worse ability to plan/organize. T Scores ≥ 65 are regarded as in the clinical range.
Executive function by report: Organization of Materials | Baseline
  Ability to organize materials will be measured using the BRIEF-2's Organization of Materials Index. Items are converted from BRIEF to BRIEF-2. Raw scores are calculated to t-scores according to the PAR BRIEF-2 manual. Higher scores means worse ability to organize materials. T Scores ≥ 65 are regarded as in the clinical range.
Executive function by report: Task-Monitor | Baseline
  The ability to task-monitor (i.e., the ability to noticing minor errors in work output) will be measured using the BRIEF-2's Task-Monitor Index. Items are converted from BRIEF to BRIEF-2. Raw scores are calculated to t-scores according to the PAR BRIEF-2 manual. Higher scores means worse ability to task-monitor. T Scores ≥ 65 are regarded as in the clinical range.
Executive function by report: Self-Monitor | Baseline
  The ability to self-monitor (i.e., the awareness of the impact of one's own behavior on other people and outcomes) will be measured using the BRIEF-2's Self-Monitor Index. Items are converted from BRIEF to BRIEF-2. Raw scores are calculated to t-scores according to the PAR BRIEF-2 manual. Higher scores means worse ability to self-monitor. T Scores ≥ 65 are regarded as in the clinical range.
Overall executive function by report | Baseline
  The childrens' overall executive function will be measured using the BRIEF-2's Global Executive Composite (Total Score). Items are converted from BRIEF to BRIEF-2. Raw scores are calculated to t-scores according to the PAR BRIEF-2 manual. Higher scores means worse executive function. T Scores ≥ 65 are regarded as in the clinical range.
Executive function by report: Behavior Regulation | Baseline
  The childrens' ability to regulate and monitor their behavior effectively will be measured using the BRIEF-2's Behavior Regulation Index (BRI). BRIEF scores are converted to BRIEF-2 scores as BRIEF-2 consists of no new items. Raw scores are calculated to T Scores according to the PAR BRIEF-2 scoring manual. Higher scores means worse behavior regulation. T Scores ≥ 65 are regarded as in the clinical range.
Executive function by report: Emotion Regulation | Baseline
  The childrens' ability to regulate their emotions will be measured using the BRIEF-2's Emotion Regulation Index (ERI). BRIEF scores are converted to BRIEF-2 scores as BRIEF-2 consists of no new items. Raw scores are calculated to T Scores according to the PAR BRIEF-2 scoring manual. Higher scores means worse emotion regulation. T Scores ≥ 65 are regarded as in the clinical range.
Executive function by report: Cognitive Regulation | Baseline
  The childrens' ability to control and manage cognitive processes and problem solve effectively will be measured using the BRIEF-2's Cognitive Regulation Index (CRI). BRIEF scores are converted to BRIEF-2 scores as BRIEF-2 consists of no new items. Raw scores are calculated to T Scores according to the PAR BRIEF-2 scoring manual. Higher scores means worse cognitive regulation. T Scores ≥ 65 are regarded as in the clinical range.
Perceived Parenting Stress by report | Baseline
  Parental stress and stressful aspects of parent-child interaction will be measured by the Parenting Stress Index (PSI; parent-report).
  Results by the following PSI Indexes will be reported:
  * Child Subscale. Values: 47 (min.) - 235 (max.)
  * Parent Subscale. Values: 54 (min.) - 270 (max.)
  * Total Stress Scale. Values: 101 (min.) - 505 (max.)
  * Life Stress. Values: 0 (min.) - 79 (max.)
  Raw scores to percentiles calculation will be done using Psychological Assessment Resources' (PAR) PSI score sheet. The percentiles will be divided in the following categories: percentiles ≤ 19, percentiles between 20 and 50, percentiles between 51 and 84, and percentiles ≥ 85. Higher scores and percentiles means more distress and vice versa.
Stress Response by Cortisol levels | Baseline
  Stress Response in children and their mothers will be measured by Hair Cortisol Concentrations:
  1st cm from the scalp of children and their mothers. Indicate hair cortisol concentrations from the last month (approximately).
Attachment style in parents by report | Baseline
  The Relationships Questionnaire (RQ; Bartholomew & Horowitz, 1991) will be used to measure four attachment styles in parents. Parents are asked to rate their degree of correspondence (7-point scale) to each attachment prototype described in RQ. The minimum value is 1 ("Disagree strongly") and the maximum value is 7 ("Agree strongly") which indicate how well or poorly each attachment style corresponds to the parent's general relationship style.
Withdrawn and Depressed Symptoms by report | Baseline
  The Syndrome Scale Withdrawn/Depressed from the Achenbach Systems of Empirically Based Assessment (ASEBA; Norwegian Version) for children 6-18 years by parent- and teacher-report will be used to measure withdrawn and depressed, i.e., internalizing, symptoms. Raw scores will be calculated to T-scores using a computer based program. Higher scores means worse symptom level. A t-score ≤ 64 indicates non-clinical symptoms, a t-score between 65 and 69 indicates that the child is at risk for clinical symptoms, and a t-score ≥ 70 indicates clinical symptoms.
Anxious and Depressed Symptoms by report | Baseline
  The Syndrome Scale Anxious/Depressed from the ASEBA (6-18 years by parent- and teacher-report) will be used to measure anxious and depressed, i.e., internalizing, symptoms. Raw scores will be calculated to T-scores using a computer based program. Higher scores means worse symptom level. A t-score ≤ 64 indicates non-clinical symptoms, a t-score between 65 and 69 indicates that the child is at risk for clinical symptoms, and a t-score ≥ 70 indicates clinical symptoms.
Somatic Complaints by report | Baseline
  The Syndrome Scale Somatic Complaints from the ASEBA (6-18 years by parent- and teacher-report) will be used to measure anxious and depressed, i.e., internalizing, symptoms. Raw scores will be calculated to T-scores using a computer based program. Higher scores means worse symptom level. A t-score ≤ 64 indicates non-clinical symptoms, a t-score between 65 and 69 indicates that the child is at risk for clinical symptoms, and a t-score ≥ 70 indicates clinical symptoms.
Social Problems by report | Baseline
  The Syndrome Scale Social Problems from the ASEBA (6-18 years by parent- and teacher-report) will be used to measure social problems. Raw scores will be calculated to T-scores using a computer based program. Higher scores means worse symptom level. A t-score ≤ 64 indicates non-clinical social problems, a t-score between 65 and 69 indicates that the child is at risk for clinical social problems, and a t-score ≥ 70 indicates clinical social problems.
Thought Problems by report | Baseline
  The Syndrome Scale Thought Problems from the ASEBA (6-18 years by parent- and teacher-report) will be used to measure thought problems. Raw scores will be calculated to T-scores using a computer based program. Higher scores means worse symptom level. A t-score ≤ 64 indicates non-clinical thought problems, a t-score between 65 and 69 indicates that the child is at risk for clinical thought problems, and a t-score ≥ 70 indicates clinical thought problems.
Attention Problems by report | Baseline
  The Syndrome Scale Attention Problems from the ASEBA (6-18 years by parent- and teacher-report) will be used to measure attention problems. Raw scores will be calculated to T-scores using a computer based program. Higher scores means worse symptom level. A t-score ≤ 64 indicates non-clinical attention problems, a t-score between 65 and 69 indicates that the child is at risk for clinical attention problems, and a t-score ≥ 70 indicates clinical attention problems.
Rule-Breaking Behavior by report | Baseline
  The Syndrome Scale Rule-Breaking Behavior from the ASEBA (6-18 years by parent- and teacher-report) will be used to measure rule-breaking behavior. Raw scores will be calculated to T-scores using a computer based program. Higher scores means worse symptom level. A t-score ≤ 64 indicates non-clinical rule-breaking behavior, a t-score between 65 and 69 indicates that the child is at risk for clinical rule-breaking behavior, and a t-score ≥ 70 indicates clinical rule-breaking behavior.
Aggressive Behavior by report | Baseline
  The Syndrome Scale Aggressive Behavior from the ASEBA (6-18 years by parent- and teacher-report) will be used to measure aggressive behavior. Raw scores will be calculated to T-scores using a computer based program. Higher scores means worse symptom level. A t-score ≤ 64 indicates non-clinical aggressive behavior, a t-score between 65 and 69 indicates that the child is at risk for clinical aggressive behavior, and a t-score ≥ 70 indicates clinical aggressive behavior.
Internalizing problems by report | Baseline
  Internalizing problems will be assessed with parent- and teacher-report using the ASEBA for children 6-18 years. The Internalizing Problems Scale Score combine the the following Syndrome Scales Scores: Anxious/Depressed, Withdrawn/Depressed, and Somatic Complaints. Higher scores means worse symptom level. T-scores from the Internalizing Problems Scale will be calculated using a computer based program. A t-score ≤ 59 indicates non-clinical symptoms, a t-score between 60 and 64 indicates that the child is at risk for problem behaviors, and a t-score ≥ 65 indicates clinical symptoms.
Externalizing problems by report | Baseline
  Externalizing problems will be assessed with parent- and teacher-report using the ASEBA for children 6-18 years. The Externalizing Problems Scale Score combine the the following Syndrome Scales Scores: Rule-Breaking Behavior and Aggressive Behavior. T-scores from the Externalizing Problems Scale will be calculated using a computer based program. Higher scores means worse symptom level. A t-score ≤ 59 indicates non-clinical symptoms, a t-score between 60 and 64 indicates that the child is at risk for problem behaviors, and a t-score ≥ 65 indicates clinical symptoms.
Total behavior and emotional problems by report | Baseline
  Total behavior and emotional problems will be assessed with parent- and teacher-report using the ASEBA for children 6-18 years. The Total Problems Scale Score combine the total Syndrome Scales Scores. This includes the following syndrome scales in addition to those included in the Internalizing and Externalizing Problems Scales: Social Problems, Thought Problems, and Attention Problems. T-scores from the Total Problems Scale will be calculated using a computer based program. Higher scores means worse symptom level. A t-score ≤ 59 indicates non-clinical symptoms, a t-score between 60 and 64 indicates that the child is at risk for problem behaviors, and a t-score ≥ 65 indicates clinical symptoms.
Affective Symptoms by report | Baseline
  The DSM-Oriented Scale Affective Problems of the ASEBA for children 6-18 years by parent- and teacher-report will be used to measure affective symptoms. Raw scores will be calculated to T-scores using a computer based program. Higher scores means worse symptom level. A t-score ≤ 64 indicates non-clinical symptoms, a t-score between 65 and 69 indicates that the child is at risk for clinical symptoms, and a t-score ≥ 70 indicates clinical symptoms. The DSM-5 oriented symptoms by ASEBA includes:
Anxiety Symptoms by report | Baseline
  The DSM-Oriented Scale Anxiety Problems of the ASEBA (6-18 years by parent- and teacher-report) will be used to measure anxiety symptoms. Raw scores will be calculated to T-scores using a computer based program. Higher scores means worse symptom level. A t-score ≤ 64 indicates non-clinical symptoms, a t-score between 65 and 69 indicates that the child is at risk for clinical symptoms, and a t-score ≥ 70 indicates clinical symptoms.
Somatic Problems by report | Baseline
  The DSM-Oriented Scale Somatic Problems of the ASEBA (6-18 years by parent- and teacher-report) will be used to measure somatic problems. Raw scores will be calculated to T-scores using a computer based program. Higher scores means worse symptom level. A t-score ≤ 64 indicates non-clinical symptoms, a t-score between 65 and 69 indicates that the child is at risk for clinical symptoms, and a t-score ≥ 70 indicates clinical symptoms.
Attention Deficit/Hyperactivity Symptoms by report | Baseline
  The DSM-Oriented Scale Attention Deficit/Hyperactivity Problems of the ASEBA (6-18 years by parent- and teacher-report) will be used to measure attention deficit/hyperactivity symptoms. Raw scores will be calculated to T-scores using a computer based program. Higher scores means worse symptom level. A t-score ≤ 64 indicates non-clinical symptoms, a t-score between 65 and 69 indicates that the child is at risk for clinical symptoms, and a t-score ≥ 70 indicates clinical symptoms.
Oppositional Defiant Symptoms by report | Baseline
  The DSM-Oriented Scale Oppositional Defiant Problems of the ASEBA (6-18 years by parent- and teacher-report) will be used to measure oppositional defiant Symptoms. Raw scores will be calculated to T-scores using a computer based program. Higher scores means worse symptom level. A t-score ≤ 64 indicates non-clinical symptoms, a t-score between 65 and 69 indicates that the child is at risk for clinical symptoms, and a t-score ≥ 70 indicates clinical symptoms.
Conduct Problems by report | Baseline
  The DSM-Oriented Scale Conduct Problems of the ASEBA (6-18 years by parent- and teacher-report) will be used to measure conduct problems. Raw scores will be calculated to T-scores using a computer based program. Higher scores means worse symptom level. A t-score ≤ 64 indicates non-clinical symptoms, a t-score between 65 and 69 indicates that the child is at risk for clinical symptoms, and a t-score ≥ 70 indicates clinical symptoms.
Irritability by report | Baseline
  The following items of the ASEBA for children 6-18 years by parent- and teacher report will be used to measure irritability symptoms on a continous scale: 86. Stubborn, Sullen, or Irritable, 87. Sudden mood changes, and 95. Temper tantrums or hot temper. Each item is rated on the same 0-1-2 Likert scale: 0 = Not True, 1 = Somewhat or Sometimes True, 2 = Very True or Often True. Minimum value is 0 and Maximum value is 6. Higher scores means more irritability and vice versa.
Dysregulation by report | Baseline
  Degree of emotional and behavioral dysregulation is computed by summing up the T-scores for the syndrome scales Anxiety/Depression, Attention Problems, and Aggression Problems (AAA profile) in ASEBA. Higher t-score means higher degree of dysregulation and vice versa. T scores equal to or above 210 means severe dysregulation.
Global Functioning | Baseline
  Children's Global Assessment Scale is a numeric scale (ranging from 1 to 100) measuring the general functioning of children. Higher scores means better functioning and vice versa.
Follow-up (6 months): Disruptive Mood Dysregulation Disorder | Follow-up at 6 months
  Children meeting criteria for Disruptive Mood Dysregulation Disorder (DMDD) at baseline will be examined after 6 months using the K-SADS screening and additional interview for DMDD to check if they still meet criteria for DMDD.
Follow-up (12 months): Diagnosis | Follow-up at 12 months
  All participants will be examined after 12 months using the K-SADS to check if they still meet the criteria for a diagnosis.
Follow-up (12 months): Symptoms | Follow-up at 12 months
  The same scales from the ASEBA as examined at baseline will be used similarly to measure symptom levels after 12 months.
Affective Interpretation Bias | Baseline
  Items examination of NEPSY-2 Affect Recognition targeting face-emotion interpretation bias.

CONTACTS AND LOCATIONS:
Overall Officials: Pål Zeiner, PhD, Study Director — Head of Child Psychiatric Research at Oslo University Hospital
Locations (2):
- Norway (2):
  - Department of Child and Adolescent Psychiatry, Oslo University Hospital, Oslo
  - Nic Waals Institute, Lovisenberg Hospital, Oslo

IPD SHARING:
Plan to Share IPD: Undecided
The data are on patients. We need to decide whether or not anonymous data can be shared with other researchers.

REFERENCES:
- See also: Regional Committees for Medical and Health Research Ethics Approval — https://helseforskning.etikkom.no/prosjekterirek/prosjektregister/prosjekt?p_document_id=811267&p_parent_id=816252&_ikbLanguageCode=n